CLINICAL TRIAL: NCT00406484
Title: Brief Introductory Therapy for Opioid Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0607001647; 2R01DA013108-04 (NIH)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Opiate Dependence; HIV Infections
Keywords: Methadone; Counseling; HIV risk reduction; HIV Seronegativity
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Behavioral Drug and HIV Risk Reduction Counseling (BDRC)
  Interventions: Behavioral: BDRC
- 2 (Active Comparator): Standard drug counseling
  Interventions: Behavioral: Standard drug counseling

INTERVENTIONS:
Behavioral: Standard drug counseling — Individual drug counseling
  Arms: 2
Behavioral: BDRC — Behavioral Drug and HIV Risk Reduction Counseling, individual once or twice weekly sessions
  Arms: 1

SUMMARY:
A randomized clinical trial to compare the efficacy of Behavioral Drug and HIV Risk Reduction Counseling (BDRC) and standard methadone drug counseling.

DETAILED DESCRIPTION:
The proposed study plans to compare the efficacy of behavioral drug and HIV risk reduction counseling (BDRC) to low intensity methadone counseling during methadone maintenance treatment. In selecting BDRC, we were guided by several considerations, including its acceptability, suitability, feasibility, potential efficacy, and potential for rapid and widespread dissemination in the U.S. and elsewhere. BDRC was developed to be delivered by regular drug counselors, so that it would be relatively easy to disseminate this counseling if it is found efficacious. BDRC combines behavioral contracting with an Information-Motivation-Behavioral Skills (IMB) model for reducing HIV risk behaviors and illicit drug use that is grounded in social cognitive theory and supported by empirical findings in a number of studies and populations. The more intensive HIV risk reduction interventions provided in BDRC, including personalized assessment of risk (i.e., identification of personal, social and environmental factors associated with risky behaviors) and education and training in skill-building and self-control, may lead to greater reductions in both drug- and sex-related HIV risk behaviors than the more limited, brief counseling provided in LIMC, as supported by findings of a recent clinical trial with methadone maintained patients and a meta-analysis regarding the effectiveness of HIV risk reduction interventions during drug abuse treatment. BDRC emphasizes a medical model of treatment for drug dependence and is highly complementary to and compatible with regular methadone maintenance treatment.

Because early abstinence achievement is associated with longer term treatment success, BDRC uses short-term behavioral contracts to help the patient achieve an initial period of abstinence, take maintenance medications regularly and as prescribed, activate the patient behaviorally, and reduce behaviors associated with HIV transmission. The accomplishment of specific, short-term behavioral goals early in treatment promotes the patient's experience of therapeutic success and counters the patient's belief that his/her actions will not lead to success in accomplishing goals. Short-term behavioral goals target a limited number of domains, including achieving an initial period of abstinence, increasing activities (primarily vocational, social or recreational) that are not related to drug use, and reducing HIV risk behaviors (e.g., fostering consistent condom use, avoiding casual sexual encounters, avoiding IDU or needle or equipment sharing). BDRC teaches cognitive and behavioral strategies for promoting behavioral change, including identifying antecedents of drug use, needle sharing, and high risk sexual behaviors, and learning strategies to avoid high risk situations or cope without engaging in these behaviors. Skill building exercises (e.g., regarding condom use) are used within sessions to learn and practice new skills, and patients are encouraged to practice these skills outside the session in their natural environment. Based on recent findings from research in cognitive and social psychology on message framing, the treatment also emphasizes the positive consequences of behavioral change (e.g., the benefits of not using drugs or of maintaining a steady relationship vs. the dangers associated with continued use or sex with multiple partners). Counselors are trained to acknowledge the patient's efforts to change-even partial accomplishments of goals are praised--rather than to focus on the patient's failures, which is often perceived as criticism. Recognition of accomplishments and positively framed messages generally evoke positive affect, which is often generalized and ascribed to the behavior in question, thus resulting in greater adherence to recommendations. An emphasis on recognition of accomplishments and positively-framed advice helps patients to build self-esteem and the sense that they can change their lives for the better.

Substance abuse is thought to be associated with a range of memory and executive function (EFs) deficits, but the majority of research support for this hypothesis comes from research on alcohol and stimulant related disorders. The evidence of long-term cognitive deficits in chronic opiate users is limited, nonetheless most consistently it suggests that EFs may be affected by chronic opiate use. Because BDRC incorporates many cognitive behavioral therapeutic techniques, includes educational and learning components and aims at improving decision making skills of the patients, we plan to evaluate a broad range of memory and executive functions of patients enrolled in the proposed study in order to identify common EFs impairments, evaluate if such impairments interfere with treatment efficacy, and if additional treatment components are necessary and can be devised in order to improve treatment efficacy for patients with cognitive impairments. We also plan to evaluate if cognitive performance improves during methadone maintenance treatment when combined with BDRC and evaluate whether presence or absence of impairments are associated with differential effects of treatments.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence

Exclusion Criteria:

* suicide or homicide risk
* psychiatric disorder requiring medication treatment
* life threatening or unstable medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum number of consecutive weeks of opiate abstinence achieved during treatment | 12 weeks
Overall proportion of opiate negative urines tests in each treatment group | 12 weeks
Reduction in HIV risk behaviors | 12 weeks

SECONDARY OUTCOMES:
Improvements in social, employment, legal, medical and psychiatric functioning | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marek C Chawarski, Ph.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Methadone Research Unit, The APT Foundation, Inc., New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut